CLINICAL TRIAL: NCT03530592
Title: Seated Ankle Robot for Foot Drop in Aging and Disabled Populations: A Demonstration Project
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baltimore VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Charlene Elaine Hafer-Macko, Associate Professor of Neurology, Baltimore VA Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-68734
Record Dates: First submitted 2018-04-10; First posted 2018-05-21 (Actual); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Peripheral Nervous System Diseases; Gait Disorders, Neurologic; Foot Drop; Mobility Limitation
MeSH Terms: conditions — Peripheral Nervous System Diseases; Gait Disorders, Neurologic; Peroneal Neuropathies; Mobility Limitation

STUDY DESIGN:
Intervention Model Description: Seated Ankle Robot Taining
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Seated Ankle Robot Training (Experimental)
  Interventions: Device: Seated Ankle Robot Training

INTERVENTIONS:
Device: Seated Ankle Robot Training — This intervention employs the use of an adaptive ankle robot control system over a 6-week intervention period.

SUMMARY:
The purpose of this research study is to test the utility of an ankle robot in people with ankle weakness and foot drop from a peripheral nervous system injury due to neuromuscular or orthopedic injury.

DETAILED DESCRIPTION:
Many individuals with central nervous system (CNS) injuries (e.g., a stroke) or peripheral nervous system (PNS) injuries (e.g., peroneal nerve injury, neuropathy, radiculopathy, and/or musculoskeletal injury) that affect their ankle movement have residual impairments that affect their walking and balance. These impairments include the disability "foot drop," which increases the risk for falling.

This study will focus on PNS injuries that cause foot drop.

Current therapy to address foot drop is limited primarily to the use of ankle foot orthoses (braces) that help keep the foot from hitting the ground to prevent falling. Also, some individuals with foot drop use functional electrical stimulation to the leg nerve to lift the foot. Regardless, none of these, or other existing, methods to address foot drop cures or even improves significantly the underlying neurological deficit behind this disability. Braces improve walking safety only while they are worn, and functional electrical stimulation does not work when it is turned off, or when the nerve has been severely damaged. Thus, the increased fall risk due to foot drop is generally considered life-long and incurable.

The investigators have developed a shoe-interfaced ankle robot with an adaptive control system, to assist an individual with ankle movement only as needed. Data from the investigators' previous studies on foot drop due to stroke show great promise for this ankle robot as a new rehabilitation tool for invididuals with foot drop. The investigators would like to utilize our findings from these stroke studies in learning how they can be used for PNS-related foot drop.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, aged 18 to 88 years
2. Chronic foot drop and ankle weakness in one leg from a peripheral nervous system injury due to a neuromuscular or orthopedic injury
3. Ability to walk 10 meters and arise from a chair with no human assistance (but usage of usual assistive device[s] is permitted)

Exclusion Criteria:

1. Medical history that would preclude participation in low-intensity seated robotic-assisted rehabilitation
2. Current participation in orthopedic or rehabilitation medical programs
3. Active deep venous thrombosis
4. Distal paretic leg skin lesions, infections, or soft tissue inflammation

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-06-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Ankle dorsiflexion-plantarflexion range of motion | Change from baseline to: post-6 weeks of training, and 6 weeks after completion of training
  degrees
Ankle inversion-eversion range of motion | Change from baseline to: post-6 weeks of training, and 6 weeks after completion of training
  degrees
Gait velocity during self-selected overground walking | Change from baseline to: post-6 weeks of training, and 6 weeks after completion of training
  cm/sec
Postural sway areas during quiet standing | Change from baseline to: post-6 weeks of training, and 6 weeks after completion of training
  cm^2; extent of postural deviations to assess static postural control
Ratio of asymmetric loading in quiet standing | Change from baseline to: post-6 weeks of training, and 6 weeks after completion of training
  ratio of Newtons of force per leg while standing quietly
Push-off forces during gait initiation | Change from baseline to: post-6 weeks of training, and 6 weeks after completion of training
  Newtons; magnitude of forward ground reaction forces.

CONTACTS AND LOCATIONS:
Overall Officials: Charlene E. Hafer-Macko, M.D., Principal Investigator — Baltimore VA Medical Center
Locations (1):
- Baltimore VA Medical Center, Baltimore, Maryland, United States